CLINICAL TRIAL: NCT02199743
Title: Lurasidone Effects on Tissue Glutamate in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Carol A. Tamminga, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 032012-053
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective; cognition; lurasidone; Latuda
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Lurasidone Hydrochloride; Haloperidol; Perphenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lurasidone (Active Comparator): Lurasidone 40mg po qhs with food x 1 week; Lurasidone 80mg po qhs with food x 3 weeks
  Interventions: Drug: Lurasidone; Drug: Haloperidol; Drug: Perphenazine
- Haloperidol (Active Comparator): Haloperidol 4mg po qhs with food x 1 week; Haloperidol 8mg po qhs with food x 3 weeks.
  Interventions: Drug: Lurasidone; Drug: Haloperidol; Drug: Perphenazine
- Perphenazine (Active Comparator): Perphenazine 16mg po qhs with food x 1 week; Perphenazine 32mg po qhs with food x 3 weeks.
  Interventions: Drug: Lurasidone; Drug: Haloperidol; Drug: Perphenazine

INTERVENTIONS:
Drug: Lurasidone — Compare to haloperidol and perphenazine
  Other Names: Latuda
Drug: Haloperidol — Compare to lurasidone
  Other Names: Haldol
Drug: Perphenazine — Compare to lurasidone
  Other Names: Trilafon

SUMMARY:
24 individuals with schizophrenia or schizoaffective disorders, who are currently considered stable, will be recruited, screened for entry criteria into a blinded study with a 4-week randomization to either lurasidone, haloperidol, or perphenazine to examine glutamate-related outcomes with lurasidone as compared to haloperidol and perphenazine.

DETAILED DESCRIPTION:
At study start all volunteers will be discontinued from their current antipsychotic drug (APD) and switched to haloperidol 4mg for 5 days. At the end of this discontinuation period, all baseline symptom ratings and cognition testing will be done, as well as the baseline imaging procedures. At the end of the baseline procedures, volunteers will be blindly randomized, either to lurasidone at 40mg (N=12), or to haloperidol at 4mg/d or perphenazine at 16mg/d (N=12). Doses will increase to 80mg/d lurasidone, 8 mg/d haloperidol, or 32 mg/d of perphenazine at the beginning of week two. Dose should be stable for the last 3 weeks of treatment unless side effects are prominent, then the dose can be decreased to 40 lurasidone/4 haloperidol/16 perphenazine mg/d for optimal clinical management. The randomization strategy will be designed and implemented by the research pharmacist in four blocks of six volunteers; drug will be dispensed by the research pharmacy according to the randomization schedule. The randomization will be followed by a four week treatment period at optimal dose levels. On the last two days of the 4 week stable dosing period, the specified glutamate outcome measures will be completed (neuroimaging and cognitive testing) along with all the symptom outcome measures, testing for drug plasma levels, and usual blood safety measures. Patients will be seen weekly for clinical evaluation; suicidality will be monitored weekly. All medications other than study drugs will be discontinued, as much as possible, for the 24-48 hr assessment period. After the evaluation phase, patients will be cross-titrated back to their original treatment medication and dosing.

This design will generate outcomes from 12 patients on lurasidone vs. 12 patients on haloperidol/ perphenazine.

ELIGIBILITY:
Inclusion Criteria:

* Subject at least 18 years old
* Subject meets criteria diagnosis of schizophrenia or schizoaffective disorder.
* Subject is not pregnant and is not planning pregnancy within the projected duration of the study.
* Female subject who is of reproductive potential agrees to remain abstinent or use adequate and reliable contraception throughout the study
* Subject is in good physical health on the basis of medical history, physical examination, and laboratory screening.
* Eyesight corrected to 20-40 or better
* Able to read, speak, and understand English*

Exclusion Criteria:

* Any medications being used as mood stabilizers (i.e., anticonvulsants)
* Subject currently has a clinically significant medical condition(s) that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study.
* Subject demonstrates evidence of acute/chronic hepatitis which is clinically significant
* Subject has a history of malignancy < 5 years prior
* Subject has a history of neuroleptic malignant syndrome (NMS).
* Subject has a history of alcohol or substance abuse within 3 months prior to screening or alcohol or substance dependence within 12 months prior to screening
* Subject tests positive for drugs of abuse at screening. In the event a subject tests positive for cannabis, the investigator will evaluate the subject's ability to abstain from cannabis during the study.
* Subjects diagnosed with type 1 diabetes
* Subject has a prolactin concentration > 200 ng/mL at screening
* Subject has a history or presence of abnormal ECG which is clinically significant
* Subject has a history of hypersensitivity to more than two distinct chemical classes of drug (e.g., sulfas and penicillins).
* Subjects have received depot neuroleptics within 12 weeks prior to randomization.
* Subject has a history of treatment with clozapine for refractory psychosis and/or subject has been treated with clozapine within 4 months of randomization.
* Subject does not have a stable residence for the 3 months prior to randomization.
* Subject requires treatment with any potent CYP3A4 inhibitors or inducers during the study.
* Subject has received electroconvulsive therapy (ECT) within 90 days prior to
* Subject has been randomized in a prior clinical trial of lurasidone.
* History of serious head injury with unconsciousness for >30 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Tamminga, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Storman D, Koperny M, Styczen K, Datka W, Jaeschke RR. Lurasidone versus typical antipsychotics for schizophrenia. Cochrane Database Syst Rev. 2025 Jan 20;1(1):CD012429. doi: 10.1002/14651858.CD012429.pub2. PMID 39831535
- See also: Tamminga Lab and Clinic Website — http://www.utsouthwestern.edu/labs/schizophrenia/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 individuals initially signed the Informed Consent and began the Screening procedures. Only 24 made it to Randomization, with only 22 making it to the end of the study. Generally participants were discontinued because they were lost to follow-up (which requires 3 telephone calls and a letter) and irregular labs that were exclusionary.
Groups:
- Lurasidone: Lurasidone 40mg po qhs with food x 1 week; Lurasidone 80mg po qhs with food x 3 weeks
  This group was compared to the "Non-Lurasidone" group (with both haloperidol and perphenazine together) in the final analysis.
- Non-Lurasidone: Haloperidol 4mg po qhs with food x 1 week; Haloperidol 8mg po qhs with food x 3 weeks.
  OR Perphenazine 8mg po qhs with food x 1 week; Perphenazine 32mg po qhs with food x 3 weeks.
  Each of these drug groups were treated individually in the study but grouped together into a "Non-Lurasidone" group for analysis.
Period: Overall Study
Arm/Group | Lurasidone | Non-Lurasidone
Started | 14 | 10
Completed | 14 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Lurasidone: Lurasidone 40mg po qhs with food x 1 week; Lurasidone 80mg po qhs with food x 3 weeks
  Compare to haloperidol and perphenazine groups combined to lurasidone group.
- Non-Lurasidone: Haloperidol 4mg po qhs with food x 1 week; Haloperidol 8mg po qhs with food x 3 weeks.
  OR Perphenazine 16mg po qhs with food x 1 week; Perphenazine 32mg po qhs with food x 3 weeks.
  Compare haloperidol and perphenazine groups combined to lurasidone.
- Total: Total of all reporting groups
Arm/Group | Lurasidone | Non-Lurasidone | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 51 [34 to 60] | 46 [36 to 58] | 49 [34 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Glutamate Levels
Description: Mean values of cerebral glutamate levels was measured by high resolution 3T magnetic resonance spectroscopy (MRS) in the anterior cingulate cortex (ACC). Data were acquired from the dorsal anterior cingulate cortex (ACC) using single voxel localized PRESS (TE1, TE2) = (32, 65) ms with an 8-channel head coil in a 3T whole-body scanner (Philips Medical Systems). Voxel size was 30x20x15 mm3 (9 mL) and were placed over the bilateral anterior cingulate cortex (ACC). All values are normalized to water.
  More negative values represent less cerebral glutamate levels.
Time Frame: Baseline and 4 weeks
Population: Of the original 22 participants, only 15 have both Baseline and Week 4 scans to compare.
Measure: Mean (Standard Deviation); unit: relative unit (RU as compared to water)
Arm/Group | Lurasidone | Non-Lurasidone
Number analyzed (Participants) | 8 | 7
relative unit (RU as compared to water)
  Baseline (week 0) | -1.434662171 (0.741430931) | -1.933853656 (1.005387144)
  week 4 | -1.412294235 (0.952600355) | -1.838991525 (1.20411535)

2. Secondary Outcome: Brief Assessments of Cognition in Schizophrenia Scores (BACS)
Description: Mean of cognition was assessed by BACS, which measures neurocognitive function in schizophrenia. BACs is a validated, composite measure of cognition which is used in schizophrenia. It is composed of Verbal memory (range: 0-75), Working memory (range: 0-28), Motor speed (range: 0-100), Verbal Fluency (number of words generated), Information processing (range: 0-110) and Executive functions (range: 0-22).
  Higher z-scores indicate a better performance and outcome. BACS composite score are represented as z-scores which can be positive or negative. There is no minimum or maximum as this is a continuous measure.
Time Frame: Baseline and 4 weeks
Population: Of the original 22 participants, only 15 have both Baseline and Week 4 to compare.
Measure: Mean (Standard Deviation); unit: BACS composite score (z score)
Arm/Group | Lurasidone | Non-Lurasidone
Number analyzed (Participants) | 8 | 7
BACS composite score (z score)
  Baseline (week 0) | -1.596573107 (0.929835487) | -1.933853656 (1.005387144)
  week 4 | -2.002433521 (1.596431421) | -1.500292967 (1.477111055)

ADVERSE EVENTS:
Groups:
- Lurasidone (LUR): Lurasidone 40mg po qhs with food x 1 week; Lurasidone 80mg po qhs with food x 3 weeks
  Compare lurasidone (LUR) group to haloperidol and perphenazine (NONLUR) group
- NONLUR: Haloperidol 4mg po qhs with food x 1 week; Haloperidol 8mg po qhs with food x 3 weeks.
  OR Perphenazine 16mg po qhs with food x 1 week; Perphenazine 32mg po qhs with food x 3 weeks.
  Compare haloperidol and perphenazine (NONLUR) group to lurasidone (LUR) group.
Arm/Group | Lurasidone (LUR) | NONLUR
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/8
Other Adverse Events (participants affected / at risk) | 3/14 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (LUR) (N=14) | NONLUR (N=8)
diabetes mellitus (Endocrine disorders) | 1 (1) | 0 (0) — Participant was monitoring glucose on his own with his PCP. Became sick with pneumonia and had his glucose increase to 315 at time of visit to ER. Was hospitalized for ~1 week. Started on medication for hypertension and insulin for DMII.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (LUR) (N=14) | NONLUR (N=8)
Sedation (Psychiatric disorders) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Insomnia (General disorders) | 3 (3) | 0 (0)
Restlessness (General disorders) | 0 (0) | 3 (3)
Stiffness in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No